CLINICAL TRIAL: NCT03598387
Title: The Study of Safety, Feasibility and Efficacy of Automated Peritoneal Dialysis in Acute Kidney Injury as Compared With Intermittent Hemodialysis, a Multi-center Non-blind Randomized Controlled Trial
Brief Title: Automated Peritoneal Dialysis Versus Intermittent Hemodialysis in Acute Kidney Injury
Acronym: SAFE-APD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Limeng Chen (Other)
Collaborators: First Hospital of China Medical University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Beijing Anzhen Hospital (Other); Xiangya Hospital of Central South University (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor-Investigator, Limeng Chen, Professor of Medicine, Associate Chief of Nephrology Division, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APD-AKI
Record Dates: First submitted 2018-06-10; First posted 2018-07-26 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; automated peritoneal dialysis; intermittent hemodialysis; renal recovery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Subjects eligible for this study will be randomized into APD group and IHD group. In APD group, subjects will receive PD catheter placement and subsequent APD treatment. In IHD group, subjects will receive un-tunneled hemodialysis catheter placement and subsequent hemodialysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APD group (Experimental): Subjects will receive PD catheter placement and subsequent automated peritoneal dialysis treatment.
  Interventions: Other: Automated peritoneal dialysis
- IHD group (Active Comparator): Subjects will receive un-tunneled hemodialysis catheter placement and subsequent intermittent hemodialysis.
  Interventions: Other: Intermittent hemodialysis

INTERVENTIONS:
Other: Automated peritoneal dialysis — The prescription of automated peritoneal dialysis:
  * The first 48-72 hours dose: 0.8-2.0 liter exchange with 1-2 hour-cycle (8-36 liters per day); After initial 48-72 hours, 1.0-2.5L exchange with 2-6 hour-cycle (at least 8 liters per day), if the acidosis, hyperkalemia and pulmonary edema are corrected.
  * The minimal target weekly Kt/V is 2.1-3.5/W.
  Arms: APD group
Other: Intermittent hemodialysis — Intermittent hemodialysis will be performed 3-4h of each session and 2-5 times per week. The prescription will be adjusted based on patients' conditions to ensure spKT/V≥1.3.
  Arms: IHD group

SUMMARY:
This is a multi-center randomized clinical trial study. The purpose of this study is to examine safety, feasibility and efficacy of automated peritoneal dialysis as compared with intermittent hemodialysis for AKI patients with indications for dialysis.

DETAILED DESCRIPTION:
The incidence of acute kidney injury (AKI) is rapidly increasing worldwide. This is a common and devastating disorder, especially in critical illnesses, affecting 5-8% of all hospitalized patients and up to 30% of those in intensive care units, with high mortality. About 50-80% critical patients with AKI needed dialysis treatment. Intermittent hemodialysis (IHD) might be the most-commonly modalities applied in AKI patients requiring dialysis. However, no data of randomized study concerning renal recovery and treatment efficiency of AKI patients treated with APD is available in Chinese adult patients. This study is a 2-armed randomized controlled non-blind non-inferior trial to explore the feasibility, efficacy, and safety of APD in AKI patients as compared with intermittent hemodialysis. Base on the sample size estimation, 100 subjects (n=50 in each arm) should be enrolled in this study. The primary outcome is the rate of renal recovery (independence of dialysis) in the first 21days after initiation of renal replacement.

ELIGIBILITY:
Inclusion Criteria:

* AKI patients according to Acute Kidney Injury Network criteria
* Rapidly rising serum creatinine level (a sudden increase of at least 30%)
* Meeting the indications for dialysis

  * Uremia or azotemia (BUN>80 mg/dl)
  * Fluid overload (after diuretics use)
  * Electrolyte imbalance (K>5.5 mEq/L after clinical treatment)
  * Acid-base disturbance (pH<7.2 and bicarbonate<10mEq/L after clinical treatment)

Exclusion Criteria:

* Age under 18 years, or older than 80 years
* Urinary tract obstruction; acute interstitial nephritis or rapidly progressive glomerulonephritis needed immunoinhibitory therapy
* Previously received renal replacement therapy(RRT) of any type/presence of dialysis access during the current illness.
* Pre-existing severe chronic kidney disease (baseline serum creatinine>4mg/dl) more than 10 days prior to initiation of first RRT.
* Absolute contraindication of peritoneal dialysis such as recent abdominal surgery (<1month), multiple abdominal surgeries.
* Absolute contraindication for hemodialysis such as hemodynamic instability (systolic blood pressure <80mmHg).
* Pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of renal function recovery (independence of dialysis) | At 21 days after the initiation of dialysis
  Patients do not require dialysis, urine output>1000ml/d and progressive drop in serum creatinine(<4mg/dl) and BUN(<50mg/dl).

SECONDARY OUTCOMES:
All-cause mortality within 21 days | At 21 days after the initiation of dialysis
  The rate of all-cause of deaths at 21 days after the initiation of dialysis
All-cause mortality within 90 days | At 90 days after the initiation of dialysis
  The rate of all-cause of deaths at 90 days after the initiation of dialysis
Access related complications within 21 days | At 21 days after the initiation of dialysis
  * Infections: peritonitis (APD), catheter-related infections (IHD)
  * Mechanical complications: catheter leakage and migration (APD), catheter obstruction (IHD)
  * Exit site bleeding, pneumothorax, hernia
Access related complications within 90 days | At 90 days after the initiation of dialysis
  * Infections: peritonitis (APD), catheter-related infections (IHD)
  * Mechanical complications: catheter leakage and migration (APD), catheter obstruction (IHD)
  * Exit site bleeding, pneumothorax, hernia
Dialysis related complications within 21 days | At 21 days after the initiation of dialysis
  Hypotension, hypoglycemia, bleeding, reactions to dialyzers, etc
The percentage of participants requiring termination of primary dialysis modality | At 90 days after the initiation of dialysis
  Condtions leading to termination of primary dialysis modality, including bleeding, thromboebolism events, infections, access related complications and inadequate dialysis
Length of stay in hospital | From the time of admission to the time of discharge, up to 90 days
  The time length of stay as an inpatient
Herth Hope Index within 21 days | At 21 days after the initiation of dialysis
  Measure hope of patients using Herth Hope Index. Total possible points on the total scale is 48 points. The higher the score the higher the level of hope. To each question, strongly agree=4, agree=3, disagree=2, strongly disagree=1. Note: the scoring items need to be reversed scored in question 3 and 6.
Health Status Questionnaire (Short Form-36) score within 21 days | At 21 days after the initiation of dialysis
  Health Status Questionnaire (Short Form-36) is one of the most widely used generic measures of health-related quality of life and has been shown to discriminate between subjects with different chronic conditions and between subjects with different severity levels of the same disease.It generates 8 subscales and two summary scores. The 8 subscales are: physical functioning (Range 0-100), role limitations due to physical problems (Range 0-100), bodily pain (Range 0-100), general health perceptions (Range 0-100), vitality (Range 0-90), social functioning (Range 12.5-100), role-limitations due to emotional problems (Range 0-100), and mental health (Range 0-100). The two summary scores are the physical component summary (Range 13.6-61.9) and the mental component summary (Range 15.6-70.0). The higher the score is, the better quality of life of the patient is.
Mini-Mental State Examination (MMSE) score within 21 days | At 21 days after the initiation of dialysis
  The Mini-Mental State Examination (MMSE) is a 30-point questionnaire that is used to measure cognitive impairment. The maximum score is 30. The following three cut-off levels should be employed to classify the severity of cognitive impairment: no cognitive impairment=24-30; mild cognitive impairment=18-23; severe cognitive impairment=0-17.
Simplified Nutritional Appetite Questionnaire (SNAQ) score within 21 days | At 21 days after the initiation of dialysis
  Simplified Nutritional Appetite Questionnaire (SNAQ) ask the subject to complete answer 4 questions about the appetite. Tally the results based upon the following numerical scale: a=1, b=2, c=3, d=4, e=5. The sum of the scores for the individual items constitutes the SNAQ score. The maximum SNAQ score is 20. SNAQ score < 14 indicates significant risk of at least 5% weight loss within six months.

CONTACTS AND LOCATIONS:
Overall Officials: Limeng Chen, MD, PhD, Principal Investigator — Division of Nephrology, Peking Union Medical College Hospital
Locations (5):
- China (5):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shannxi

IPD SHARING:
Plan to Share IPD: No
To comply with laws in China, local regulations and hospital policy, IPD sharing might be restricted

REFERENCES:
- [Background] Gabriel DP, Nascimento GV, Caramori JT, Martim LC, Barretti P, Balbi AL. Peritoneal dialysis in acute renal failure. Ren Fail. 2006;28(6):451-6. doi: 10.1080/08860220600781245. PMID 16928612
- [Background] Gabriel DP, Caramori JT, Martim LC, Barretti P, Balbi AL. High volume peritoneal dialysis vs daily hemodialysis: a randomized, controlled trial in patients with acute kidney injury. Kidney Int Suppl. 2008 Apr;(108):S87-93. doi: 10.1038/sj.ki.5002608. PMID 18379555